CLINICAL TRIAL: NCT03758872
Title: USE OF ENDOCUFF SECOND GENERATION IN THE COLIC POLYPS DETECTION: HISTORIC COHORTE PROSPECTIVE COMPARATIVE
Brief Title: CUFF-assisted Colonoscopy vs Standard Colonoscopy
Acronym: CUFF-TROCADERO
Status: Completed | Type: Observational
Sponsor: Clinique du Trocadéro (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-A01397-48
Record Dates: First submitted 2018-10-26; First posted 2018-11-29 (Actual); Last update posted 2021-01-29 (Actual); Status verified 2018-10

CONDITIONS: Colonic Polyp; Colonoscopy
MeSH Terms: conditions — Colonic Polyps | interventions — Colonoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- historical comparaison whithout cuff: 517 patients included in 2017 without CUFF and 517 patients will be included in 2018 with CUFF for polyp detection
  Interventions: Diagnostic Test: cuff assisted colonoscopy(with cuff use of endocuff vision second generation)

INTERVENTIONS:
Diagnostic Test: cuff assisted colonoscopy(with cuff use of endocuff vision second generation) — this is a cohort prospective comparative, a group without cuff in 2017, 517 patient included in the retrospective phase, and in 2018, 517 patient will be included in the prospective phase with CUFF for detecting polyps
  Other Names: colonoscopy with polypectomy or mucosectomy; standard colonoscopy ( without use of endocuff vision)

SUMMARY:
The goal of this study is to evaluate the interest of second-generation Endocuff Vision (ECV) to improve Adenoma detection rate and / or Polyp detection rate in routine colonoscopy.

This is a prospective comparative cohort, on 1034 patients, 517 patients with ECV in prospective group and 517 without ECV in retrospective group

ELIGIBILITY:
Inclusion Criteria:

* Patient scheduled for total colonoscopic exploration, during the period study
* Patient over or equal to 18 years
* ASA 1, ASA 2, ASA 3
* No participation in another clinical study
* Certificate of non opposition signed

Exclusion Criteria:

* Patient under 18 years old
* ASA 4, ASA 5
* Pregnant woman
* Patient with coagulation abnormalities preventing polypectomy: prothrombin level <50%, -Platelets <50000 / mm3, effective anti-coagulation in progress, clopidogrel in progress.
* Inflammatory bowel disease
* Known colonic stenosis
* Diverticulitis less than 6 weeks old
* Patient unable to give consent or protected by law
* Opposition expressed for inclusion in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient of all participating physicians for total colonoscopic exploration over the study periods
Sampling Method: Probability Sample
Enrollment: 1034 (Actual)
Dates: Start 2018-10-25 (Actual); Primary Completion 2019-09-26 (Actual); Study Completion 2019-09-26 (Actual)

PRIMARY OUTCOMES:
detection of polyp or adenoma with cuff | during procedure

SECONDARY OUTCOMES:
POLYP DETECTION RATE | during procedure
morbidity : perforation rate | 21 DAYS AFTER PROCEDURE
CAECAL INTUBATION RATE | DURING PROCEDURE
TIME TO REACH CAECUM | DURING PROCEDURE
  SEC
WITHDRAWAL TIME | DURING PROCEDURE
  SEC

CONTACTS AND LOCATIONS:
Locations (1):
- Clinique Du Trocadero, Paris, France

IPD SHARING:
Plan to Share IPD: No